CLINICAL TRIAL: NCT02989597
Title: Single-dose Intraoperative Methadone for Early Ambulation and Sustained Pain Control in Spinal Fusion Surgery Patients
Brief Title: Intraoperative Methadone Administration for Improved Pain Control in Spinal Fusion Patients
Acronym: MAPS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to personnel loss and logistical issues the study was unable to be completed as planned.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-6985
Record Dates: First submitted 2016-12-07; First posted 2016-12-12 (Estimated); Results first posted 2023-04-25 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone; Dexamethasone; Ketamine; Remifentanil; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-operative Methadone Hydrochloride (Experimental): Patient who will be given a single dose of intra-operative methadone, and having standard care otherwise
  Interventions: Drug: Methadone Hydrochloride; Other: Standard pain regimen; Procedure: Spinal Fusion Surgery; Drug: Dexamethasone; Drug: Ketamine; Drug: Remifentanil; Drug: Sufentanil
- Control (Active Comparator): Patients administered standard of care
  Interventions: Other: Standard pain regimen; Procedure: Spinal Fusion Surgery; Drug: Dexamethasone; Drug: Ketamine; Drug: Remifentanil; Drug: Sufentanil

INTERVENTIONS:
Drug: Methadone Hydrochloride — IV administration of methadone intra-operatively for a single dose
  Arms: Intra-operative Methadone Hydrochloride
Other: Standard pain regimen — Standard medications for pain control administered after spinal surgery to be either fentanyl or morphine
Procedure: Spinal Fusion Surgery — Clinically-indicated spinal fusion surgery
Drug: Dexamethasone — Post operative swelling and pain control
Drug: Ketamine — Perioperative anesthesia medication
Drug: Remifentanil — Perioperative pain medication
Drug: Sufentanil — Perioperative pain medication

SUMMARY:
Methadone has several advantages over standard narcotic medications, especially when considering use after a typically painful surgery such as lumbar fusion. Methadone is low cost, has a long half-life, has a convenient dosing schedule, has excellent oral bioavailability, and demonstrates slow onset to withdrawal. The literature comparing methadone to more commonly used post-operative narcotics demonstrates that it manages pain better, sustains consistent plasma concentrations, decreases overall narcotic requirement, results in no additional adverse events, and is safe, even in children, across several studies. Since the standard of care is non-methadone narcotic usage to manage the significant pain of complex spinal surgery cases, it is understandable that methadone could be a desirable alternative to promote sustained pain control and early ambulation in these patients. The goal of this study is to compare the effect of a single dose of methadone administered intraoperatively in enrolled spinal fusion patients to their historical controls given fentanyl and morphine, and determine if more sustained pain control during the first few days after surgery provides a better subjective experience for the patient with less pain, which allows them to ambulate and leave the hospital sooner than patients given a standard regimen.

DETAILED DESCRIPTION:
Methadone is a synthetic opioid analgesic with agonist properties at the µ-opioid receptor binding site that has long been used as an alternative to morphine and hydromorphone in patients with severe pain. It has a diffuse bioavailability and is highly efficacious through its oral form, yet its bioavailability is heavily dependent on variability in cytochrome P450 3A4 enzyme activity, and is quite variable amongst individuals. Methadone reaches peak plasma concentrations in 2.5 to 4 hours after oral administration, has a rapid onset, has a half-life is between 20-35 hours (range 5-130 hours), and analgesia may be reported for up to 108 hours after a single dose. Additionally, methadone's NMDA (N-methyl-D-aspartate) receptor site antagonism acts to inhibit enzymes such as adenyl cyclase and their downstream production of secondary signaling molecules like cyclic AMP (adenosine monophosphate). This activity may attenuate opioid tolerance and opioid abstinence syndrome as NMDA receptor agonism has been implicated in the development of hyperalgesia, acute and chronic tolerance, and chronic pain states.

IV dosing typically ranges from 2.5mg to 10mg every 8-12 hours, with PO forms dosed at 5-20mg every 6-8 hours.

In a study of surgical patients, 40% required no additional post-operative pain control after a single 20mg iv methadone dose intra-operatively, and the 35% that did require a single additional dose required it on average 18.4±6.6 hours post-operatively. The remainder received additional non-narcotic pain medications post-operatively which were sufficient to control pain to tolerable levels.

In a series of 29 patients undergoing multilevel thoracolumbar spine surgeries with instrumentation and fusion, patients were randomized to receive either methadone (0.2mg/kg) or sufentanil infusion of 0.25µg/kg/h after a load of 0.75 µg/kg.Post-operative pain control was delivered by patient-controlled analgesia and patients were assessed by visual analogue scale for pain, opioid dose, and side effected at 1, 2, and 3 days post-operatively. Patients reported less pain in the methadone group 48 hours post-operatively, as well as used less cumulative narcotic dose than the remifentanil control group. Side effects were not significantly different between the two groups. This study however, did not evaluate post-operative functional status, ambulation, and time to discharge.

The literature comparing methadone to more commonly used post-operative narcotics demonstrates that it manages pain better, decreases narcotic requirement, results in no additional adverse events, and is safe, even in children. Since the standard of care is narcotic usage to manage the significant pain of complex spinal surgery cases, it is understandable that methadone could be a desirable therapy to promote sustained pain control and early ambulation in these patients.

The current hypothesis is that methadone use intra-operatively will result in earlier time to ambulate post op and better ability to participate with post-operative physical therapy evaluation, lower narcotic usage, and earlier discharge. It is also foreseeable that since methadone would be administered while the patient was sedated intra-operatively, it could prevent the association between the analgesia and euphoria that may result from self- or nurse-administered narcotics, such as with a patient-controlled analgesia (PCA), which could promote early tolerance or reliance. The study plans to enroll the first 30 consecutive patients who met inclusion criteria, with an end goal of 20 patients who will complete the study. Patient will be recruited in office at time of consent for surgery by the principal investigator and be scheduled to undergo 1 or 2 level lumbar decompression and fusion surgery.

The study outlined will be a prospective, positive-control, triple-blinded study in which the patient, care providers, and investigators will be unaware of the randomization of the patients. Only the anesthesiologist treating the patient during surgery will be aware of the administration of methadone or not.

On the day of surgery, the patient's pre-operative pain and functional status will be assessed, in addition to a review of the study protocols. An anesthesiologist will be assigned to the case and will administer a 0.2 mg/kg single-dose administration of methadone on incision (not to exceed 20 mg, as used in the literature) with a ketamine infusion of 4 µg/kg/min and a remifentanil infusion starting at 0.1 µg/kg/min and titrating to effect or sufentanil infusion starting with a dose of 0.3 µg/kg/hr and titrating to effect. These standard doses have been well documented and studied in the literature and will be overseen and have been approved by Board certified anesthesiologist. For lengthier procedures, there will not be re-dosing of narcotics toward the end of the procedure. The operative procedure will not be altered in any way for the purposes of this study, and is beyond the scope of this protocol, yet can be detailed as requested. The patient will be taken to the recovery room post-operative and will be put on a standard post-operative morphine PCA at a rate of 1mg per 6 minute lock-out period. Patient's narcotic usage and pain rating will be recorded at the intervals listed above and when stable from a cardiovascular standpoint, will be transition to the neurosurgery floor. Once able to bare weight, the patient will be encouraged to work with physical and occupational therapy as per standard post-operative protocol. Once the patient uses the PCA at a rate of less that once an hour, and can be managed with oral pain medications, the PCA will be removed. The remainder of their post-operative care will be according to the standard departmental protocol, and when milestones such as ambulation, voiding, and pain control are met, they will be discharged either to home, an acute care facility, or a subacute rehabilitation center. Any adverse events/reactions will be recorded and managed as normally they would be, and naloxone will be available for suspicion of narcotic overdose The subjects of this study will be compared to the historical controls in demonstrating the effect of methadone on post-operative pain, medication usage, and rehabilitation time. A goal of 30 patients will be planned to be enrolled. Other than intra-operative narcotic administration, all other portions of the intra-operative and post-operative care will remain the same as for historical patients.

The primary outcomes for the study include total narcotic dose post-operative, frequency of narcotic use, the time to first ambulation after surgery with physical therapy, length of stay, and disposition (i.e. level of rehabilitative care). Secondary outcomes include better subjective pain control, need for post-operative course of dexamethasone for post-operative/post-fusion radiculopathy or neurapraxia/neuropathy, and fusion at 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Meets age criteria, age between 18-80
* Undergoing lumbar fusion surgery, one or two spinal levels
* ASA (American Society of Anesthesiologists) grades I-III

Exclusion Criteria:

* Patient outside of age criteria
* Renal failure requiring dialysis
* Serum creatinine greater than 2.0
* Hepatic dysfunction with liver function tests greater than twice the upper limit
* Pulmonary disease requiring home oxygen therapy
* Obstructive sleep apnea
* Severe heart disease
* Allergy to methadone, morphine, or fentanyl
* Recent or distant history of opioid abuse
* Poorly managed psychiatric illness
* Known history of alcohol abuse
* Morbid obesity (body mass index > 50 kg/m2)
* Treatment with other NMDA receptor antagonists
* Prolonged QTc (corrected QT interval) on pre-operative EKG,
* Refusal or inability to sign the consent form
* Current use of HIV-1 protease inhibitors, erythromycin, ketoconazole, rifabutin, carbamazepine, phenytoin, phenobarbital, St. John's Wort, fluconazole, fluvoxamine, fluoxetine, paroxetine
* Grapefruit juice intake within the last week

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-29 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Kobets, MD, MHS, Principal Investigator — Department of Neurological Surgery, Albert Einstein School of Medicine/Montefiore Medical Center; Merritt D Kinon, MD, Principal Investigator — Department of Neurological Surgery, Albert Einstein School of Medicine/Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Background] Inturrisi CE. Pharmacology of methadone and its isomers. Minerva Anestesiol. 2005 Jul-Aug;71(7-8):435-7. PMID 16012416
- [Background] Lugo RA, Satterfield KL, Kern SE. Pharmacokinetics of methadone. J Pain Palliat Care Pharmacother. 2005;19(4):13-24. PMID 16431829
- [Background] Stemland CJ, Witte J, Colquhoun DA, Durieux ME, Langman LJ, Balireddy R, Thammishetti S, Abel MF, Anderson BJ. The pharmacokinetics of methadone in adolescents undergoing posterior spinal fusion. Paediatr Anaesth. 2013 Jan;23(1):51-7. doi: 10.1111/pan.12021. Epub 2012 Sep 14. PMID 22978825
- [Background] Sharma A, Tallchief D, Blood J, Kim T, London A, Kharasch ED. Perioperative pharmacokinetics of methadone in adolescents. Anesthesiology. 2011 Dec;115(6):1153-61. doi: 10.1097/ALN.0b013e318238fec5. PMID 22037641
- [Background] Pacreu S, Fernandez Candil J, Molto L, Carazo J, Fernandez Galinski S. The perioperative combination of methadone and ketamine reduces post-operative opioid usage compared with methadone alone. Acta Anaesthesiol Scand. 2012 Nov;56(10):1250-6. doi: 10.1111/j.1399-6576.2012.02743.x. Epub 2012 Jul 26. PMID 22834921
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Marymont JH, Shear T, Parikh KN, Patel SS, Gupta DK. Intraoperative Methadone for the Prevention of Postoperative Pain: A Randomized, Double-blinded Clinical Trial in Cardiac Surgical Patients. Anesthesiology. 2015 May;122(5):1112-22. doi: 10.1097/ALN.0000000000000633. PMID 25837528
- [Background] Jacobson L, Chabal C, Brody MC, Ward RJ, Ireton RC. Intrathecal methadone and morphine for postoperative analgesia: a comparison of the efficacy, duration, and side effects. Anesthesiology. 1989 May;70(5):742-6. doi: 10.1097/00000542-198905000-00005. PMID 2655501
- [Background] Gourlay GK, Willis RJ, Wilson PR. Postoperative pain control with methadone: influence of supplementary methadone doses and blood concentration--response relationships. Anesthesiology. 1984 Jul;61(1):19-26. PMID 6742480
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Udelsmann A, Maciel FG, Servian DC, Reis E, de Azevedo TM, Melo Mde S. Methadone and morphine during anesthesia induction for cardiac surgery. Repercussion in postoperative analgesia and prevalence of nausea and vomiting. Rev Bras Anestesiol. 2011 Nov-Dec;61(6):695-701. doi: 10.1016/S0034-7094(11)70078-2. English, Multiple languages. PMID 22063370
- [Background] Russell T, Mitchell C, Paech MJ, Pavy T. Efficacy and safety of intraoperative intravenous methadone during general anaesthesia for caesarean delivery: a retrospective case-control study. Int J Obstet Anesth. 2013 Jan;22(1):47-51. doi: 10.1016/j.ijoa.2012.10.007. Epub 2012 Dec 7. PMID 23219678

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intra-operative Methadone Hydrochloride | Control | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: The Short Form-36 (SF-36) health survey will be used as an indicator of overall health status. The SF-36 is a self-reported questionnaire which measures eight scaled scores: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Likert scales and yes/no options are used to assess function and well-being. Scales are standardized to obtain a score ranging from 0-100. Higher scores are indicative of better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Time Frame: Preoperatively
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 4 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 8 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 12 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 16 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 20 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 24 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 28 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 32 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 36 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 40 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 44 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 48 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 52 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 56 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 60 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

17. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 64 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

18. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 68 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

19. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 72 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

20. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 76 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 80 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

22. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 84 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

23. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 88 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

24. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 92 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

25. Primary Outcome: Overall Health-related Quality of Life (SF-36)
Description: as for outcome 1
Time Frame: 96 hours after surgery
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

26. Primary Outcome: Time to First Ambulation
Description: Unit: days. Assessments of patients' time to first ambulation post-operatively
Time Frame: Immediately postoperatively until ambulation, on average 3-4 days
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

27. Primary Outcome: Time to Discharge From Hospital
Description: Unit: days. Measured at patient discharge (=length of stay)
Time Frame: Immediately postoperatively until patient discharge, on average 1 week, up to 1 month
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

28. Primary Outcome: Total Narcotic Dose in the Hospital
Description: Unit: mg. Amount of narcotic used intra-operatively until study completion (patient discharge)
Time Frame: Intraoperatively until patient discharge, on average 1 week, up to 1 month
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

29. Primary Outcome: Frequency of Narcotic Usage
Description: Unit: number. Frequency of narcotics used intra-operatively until study completion (patient discharge)
Time Frame: Intraoperatively until patient discharge, on average 1 week, up to 1 month
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

30. Primary Outcome: Patient Disposition at Discharge
Description: Level of rehabilitative care deemed to be required (upon patient discharge)
Time Frame: At patient discharge, on average 1 week, up to 1 month
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Post-operative Course of Dexamethasone
Description: Binary assessment of need for post-operative course of Dexamethasone for post-operative/post-fusion radiculopathy or neurapraxia/neuropathy
Time Frame: Intraoperatively through patient discharge, on average 1 week, up to 1 month
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Assessment of Lumbar Fusion
Description: Confirmation of successful fusion of lumbar vertebrae
Time Frame: 3-6 months
Population: Data were not collected/aggregated and, as such, no data analysis was conducted.
Arm/Group | Intra-operative Methadone Hydrochloride | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Intraoperatively through patient discharge, on average 1 week, up to 1 month
Description: Risks of using any opioid narcotic, were monitored along with psychological risks, especially in opioid-naive patients. For patients in the methadone group, if the methadone intervention contributed greater than normal adverse events (>2 patients) the study would have been held from further recruitment. If this adverse event was found to have been caused by the methadone administration, the trial would have stopped.
Groups:
- Intra-operative Methadone Hydrochloride: Patients who will be given a single dose of intra-operative methadone, and having standard care otherwise
  Methadone Hydrochloride: IV administration of methadone intra-operatively for a single dose
  Standard pain regimen: Standard medications for pain control administered after spinal surgery to be either fentanyl or morphine
  Spinal Fusion Surgery: Clinically-indicated spinal fusion surgery
  Dexamethasone: Post operative swelling and pain control
  Ketamine: Perioperative anesthesia medication
  Remifentanil: Perioperative pain medication
  Sufentanil: Perioperative pain medication
Arm/Group | Intra-operative Methadone Hydrochloride | Control
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT02989597/Prot_SAP_000.pdf